CLINICAL TRIAL: NCT04754802
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of PH94B Nasal Spray for the Acute Treatment of Anxiety Induced by a Public Speaking Challenge in Adult Subjects With Social Anxiety Disorder
Brief Title: PH94B Nasal Spray for Anxiety Induced by a Public Speaking Challenge
Acronym: Palisade-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VistaGen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PH94B-CL026
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-07

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PH94B (Experimental): PH94B Nasal Spray - single treatment with 3.2 micrograms PH94B
  Interventions: Drug: PH94B Nasal Spray
- Placebo (Experimental): Placebo Nasal Spray - single treatment with placebo
  Interventions: Drug: Placebo Nasal Spray

INTERVENTIONS:
Drug: PH94B Nasal Spray — Nasal spray delivered 20 minutes before the public speaking stressor
  Arms: PH94B
Drug: Placebo Nasal Spray — Nasal spray delivered 20 minutes before the public speaking stressor
  Arms: Placebo

SUMMARY:
This Phase 3 clinical trial is designed to evaluate the efficacy, safety, and tolerability of the acute administration of 3.2 µg of PH94B to relieve symptoms of anxiety in adult subjects with social anxiety disorder (SAD) during an induced public speaking challenge.

Subject participation in the Study will last a total of 3 to 7 weeks, depending on the duration of the screening period and intervals between visits. Upon signing an informed consent, all subjects will complete Visit 1 (Screening) and enter a screening period lasting between 3 and 35 days. If subjects meet all eligibility criteria at the end of the screening period, subjects will return for Visit 2 and self-administer the nasal spray and then participate in a 5 minute public speaking challenge. During the public speaking challenge, the subject will be asked for their anxiety score, which will be recorded by a trained observer. At Visit 3, the subjects will undergo the same public speaking procedure once again as they did in Visit 2. One week after the completion of the Visit 3 public speaking challenge, the subject will come back for Visit 4 (Follow-up) that will involve a repeat of the safety and psychiatric assessments conducted at Screening.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided prior to conducting any study-specific assessment.
2. Male or female adult, 18 through 65 years of age, inclusive.
3. Current diagnosis of SAD as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, as confirmed by the Mini-International Neuropsychiatric Interview (MINI).
4. Clinician-rated Liebowitz Social Anxiety Scale (LSAS) total score ≥70 at Screening (Visit 1).
5. Clinician-rated Hamilton Depression Score 17-items total score <18 at Screening (Visit 1).
6. Women of child bearing-potential must be able to commit to the consistent and correct use of an effective method of birth control throughout the study, and must also have a negative urine pregnancy test result at both Screening (Visit 1) and Baseline (Visit 2), prior to IP administration. Effective methods of contraception include: condoms with spermicide, diaphragm with spermicide, hormonal contraceptive agents (oral, transdermal, or injectable), or implantable contraceptive devices.
7. Negative COVID-19 test either in the presence of COVID-19 symptoms or after direct exposure to someone with a positive COVID-19 test.

Exclusion Criteria:

1. Any history of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, psychosis, anorexia or bulimia, premenstrual dysphoric disorder, or obsessive-compulsive disorder. Any other current Axis I disorder, other than SAD, which is the primary focus of treatment. Note that subjects with concurrent Generalized Anxiety Disorder are eligible for the study provided that Generalized Anxiety Disorder is not the primary diagnosis.
2. Subjects who meet criteria for moderate or severe alcohol or substance use disorder within the 1 year prior to Study entry.
3. In the opinion of the investigator, the subject has a significant risk for suicidal behavior during the course of their participation in the study, or considered to be an imminent danger to themselves or others.
4. Clinically significant nasal pathology or history of significant nasal trauma, nasal surgery, anosmia, or nasal septum perforation that may have damaged the nasal chemosensory epithelium.
5. An acute or chronic condition, including an infectious illness, uncontrolled seasonal allergies at the time of the study, or significant nasal congestion that potentially could affect drug delivery to the nasal chemosensory epithelium.
6. Two or more documented failed treatment trials with a registered medication approved for SAD, taken at any time during the lifetime of the patient, whereby an adequate treatment trial is defined as that documented in the package insert for a particular drug during which the subject received an adequate medication dosage (defined as the treatment dose indicated in the package insert to obtain efficacy for that particular drug).
7. Use of any psychotropic medication within 30 days before Study entry (other than allowed medication for insomnia.
8. Concomitant use of any anxiolytics, such as benzodiazepines or unapproved treatments such as beta blockers, during the Study and within 30 days before Study entry.
9. Concomitant use of any over-the-counter, prescription product, or herbal preparation for treatment of the symptoms of anxiety or social anxiety during the Study and within 30 days before Study entry.
10. Prior participation in a clinical trial involving PH94B.
11. Women who have a positive serum or urine pregnancy test prior to IP administration.
12. Subjects with clinically significant abnormalities in hematology, blood chemistry, urinalysis, electrocardiogram, or physical examination identified at the Screening visit or Baseline visit that in the clinical judgment of the Investigator, could place the subject at undue risk, interfere with study participation, or confound the results of the study.
13. Subjects with a positive urine drug screen at either the Screening visit or Baseline visit (not including tetrahydrocannabinol).
14. Any current clinically significant and/or uncontrolled medical condition, based on medical history or as evidenced in screening assessments, such as SARS-Cov-2, HIV, cancer, stroke, congestive heart failure, uncontrolled diabetes mellitus, or any other medical condition or disease that, in the clinical judgment of the Investigator, could place the subject at undue risk, interfere with Study participation, or confound the results of the Study.
15. History of cancer or malignant tumor not in remission for at least 2 years. Basal cell skin cancers are not exclusionary.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - VistaGen Clinical Site, Los Angeles, California
  - VistaGen Clinical Site, Orange, California
  - VistaGen Clinical Site, Riverside, California
  - VistaGen Clinical Site, San Diego, California
  - VistaGen Clinical Site, San Jose, California
  - VistaGen Clinical Site, Sherman Oaks, California
  - VistaGen Clinical Sites, Fort Myers, Florida
  - VistaGen Clinical Site, Jacksonville, Florida
  - VistaGen Clinical Site, Orlando, Florida
  - VistaGen Clinical Site, Tampa, Florida
  - VistaGen Clinical Site, Chicago, Illinois
  - VistaGen Clinical Site, Watertown, Massachusetts
  - VistaGen Clinical Site, Princeton, New Jersey
  - VistaGen Clinical Site, New York, New York
  - VistaGen Clinical Site, Oklahoma City, Oklahoma
  - VistaGen Clinical Site, Allentown, Pennsylvania
  - VistaGen Clinical Site, Media, Pennsylvania
  - VistaGen Clinical Site, Houston, Texas
  - VistaGen Clinical Site, San Antonio, Texas
  - VistaGen Clinical Site, Woodstock, Vermont
  - VistaGen Clinical Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liebowitz MR, Salman E, Nicolini H, Rosenthal N, Hanover R, Monti L. Effect of an acute intranasal aerosol dose of PH94B on social and performance anxiety in women with social anxiety disorder. Am J Psychiatry. 2014 Jun;171(6):675-82. doi: 10.1176/appi.ajp.2014.12101342. PMID 24700254

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PH94B | Placebo
Started | 112 | 112
Completed | 110 | 110
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- PH94B: 3.2 micrograms PH94B intranasal spray (100 microliters to each nostril) one time
  PH94B Nasal Spray: Nasal spray delivered 20 minutes before the public speaking stressor
- Placebo: Placebo intranasal spray (100 microliters to each nostril) one time
  Placebo Nasal Spray: Nasal spray delivered 20 minutes before the public speaking stressor
- Total: Total of all reporting groups
Arm/Group | PH94B | Placebo | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 112 | 224
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (10.69) | 35.6 (11.71) | 35.3 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 73 | 150
  Male | 35 | 39 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 18 | 3 | 21
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 23 | 18 | 41
  White | 63 | 71 | 134
  More than one race | 3 | 10 | 13
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 112 | 112 | 224
Subjective Units of Distress (SUDS) score [Mean (Standard Deviation); unit: score on a scale] — The SUDS is a patient self-rated scale that is scored in the range of 0 to 100 (operationalized for participants in this study as 0=totally relaxed or no anxiety and 100=most distress or anxiety imaginable). A total of 6 SUDS scores are obtained during the 5 minute public speaking challenge. The reported SUDS score is the mean of the 6 values. If a subject does not complete 5 minutes, the mean is derived from the available scores.
  score on a scale | 77.7 (11.67) | 78.2 (12.42) | 77.95 (12.05)

OUTCOME MEASURES:

1. Primary Outcome: Subjective Units of Distress Scale (SUDS) Score
Description: The SUDS is a patient self-rated scale that is scored in the range of 0 to 100 (operationalized for participants in this study as 0=totally relaxed or no anxiety and 100=highest distress or anxiety ever felt
Time Frame: Visit 2 (Baseline; Day 0) to Visit 3 (Day 7 ± 2 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PH94B | Placebo
Number analyzed (Participants) | 112 | 112
score on a scale
  Visit 2 | 77.7 (11.67) | 78.2 (12.42)
  Visit 3 | 62.3 (19.40) | 61.3 (19.56)
Statistical Analysis 1: Comparison: PH94B vs Placebo; Test type: Superiority; p = .5063, ANCOVA; Mean Difference (Net) = 1.6, 95% CI 2-sided [-3.2 to 6.4], Standard Error of Mean 2.42

2. Secondary Outcome: Proportions (%) of CGI-I Responders in PH94B-treated and Placebo-treated Groups at the End of Visit 3 (Treatment)
Description: The CGI-I scale is a clinician-rated scale to assess illness improvement. The CGI-I scale includes one item scored from 1 (Very much less anxious) to 7 (Very much more anxious) with 4 being no change. Subjects are considered CGI-I responders with scores of 1 (Very much less anxious) or 2 (Much less anxious
Time Frame: Visit 2 (Baseline; Day 0) to Visit 3 (Day 7 ± 2 days)
Population: Although the population of analysis included n=112, one subject had no CGI-I value. No imputation was done for secondary endpoints, resulting in n=111 in the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | PH94B | Placebo
Number analyzed (Participants) | 111 | 112
Participants | 34 | 36
Statistical Analysis 1: Comparison: PH94B vs Placebo; Test type: Superiority; p = .8077, Wald Normal Approximation (Z); Wald Normal Approximation (Z) for difference between two proportions; Other = -0.015, 95% CI 2-sided [-0.137 to 0.107]

ADVERSE EVENTS:
Time Frame: 16 days
Description: One subject was randomized to PH94B but IP was neither dispensed nor administered to the subject at Visit 3
Arm/Group | PH94B | Placebo
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/112
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/112
Other Adverse Events (participants affected / at risk) | 0/111 | 0/112

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT04754802/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT04754802/SAP_001.pdf